CLINICAL TRIAL: NCT05253768
Title: Safety and Efficacy of Human Microbiota Transplantation for Overweight and Obese Type 2 Diabetes Mellitus ( SETOM ): A Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Safety and Efficacy of Human Microbiota Transplantation for Overweight and Obese Type 2 Diabetes Mellitus
Acronym: SETOM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Dongguan People's Hospital (Other Government); Shenzhen Hengsheng Hospital (Unknown); Shaoguan Qide Hospital (Unknown); Shaoguan First People's Hospital (Unknown); Zhaoqing First People's Hospital (Unknown); Suixi Hospital of Guangdong Medical University (Unknown); Shantou Central Hospital (Other); People's Hospital of Xinxing County (Unknown); Shantou Longhu People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SETOM
Record Dates: First submitted 2021-12-23; First posted 2022-02-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus; Overweight and Obesity
Keywords: Fecal Microbiota Transplantation(FMT); Type 2 Diabetes Mellitus; obesity; Weight Loss; Diabetes Mellitus; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Weight Loss; Diabetes Mellitus | interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Patients who receive a fecal microbiota transplantation via a nasointestinal tube.
  Interventions: Biological: Fecal microbiota transplant (FMT)
- placebo (Placebo Comparator): Patients who receive a placebo FMT via a nasointestinal tube.
  Interventions: Other: normal saline and glycerin/food coloring

INTERVENTIONS:
Biological: Fecal microbiota transplant (FMT) — Patients will randomized to a fecal microbiota transplantation by using a nasointestinal tube for 3 times in 4 weeks(0,2,4) without undergoing an enema before the treatment.
  The amount of FMT is 200ml at one time. Patients are given the same lifestyle guidance and nutritional advice.
  Arms: intervention
Other: normal saline and glycerin/food coloring — Patients will receive an equivalent volume of normal saline and glycerin/food coloring via a nasointestinal tube (sham transplantation) for 3 times in 4 weeks(0,2,4) without undergoing an enema before the treatment.
  The amount of placebo FMT is 200ml at one time. Patients are given the same lifestyle guidance and nutritional advice.
  Arms: placebo

SUMMARY:
The main purpose is to evaluate whether the percentage of body weight change from baseline to week 12 is higher than that in the placebo group.

In this randomized, double-blind, placebo-controlled study, 39 patients fulfilling the study criteria will be enrolled in the study. Patients will be randomized(2:1) to either FMT or placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study evaluating fecal microbiota transplantation from lean healthy donors to reduce the patients' weight. Patients wishing to participate will be evaluated whether they qualify for the study regarding the aforementioned inclusion and exclusion criteria. The details of the experiment and potential risks or discomforts involved in it will be presented, after which the patients will sign informed consent forms.

In this study, patients will be randomly assigned to the experimental group and the control group in a 2:1 ratio according to a random allocation table. The table will be formulated on the basis of the random numbers generated by SPSS.

The study will comprise of three parts:

1. Baseline - two weeks of run-in and screening period.

   * Ensure that each patient reads and signs informed consent.
   * Collect demographic data.
   * Ask about past medical history, current medical history, surgical history, allergy history, etc.
   * Ask about previous medication and combination medication.
   * Complete the FFQ questionnaire.
   * Collect information about vital signs, physical examination, BMI, ECG, conventional index and therapeutic effect index.
   * Collect 2 tubes of stool samples for fecal metagenomics sequencing and three tubes of blood samples for measuring serum metabolomics and inflammatory index (IL-6).
   * Review whether patients qualify for participate in the study according to the inclusion and exclusion criteria.
   * Dietitian will give diet, exercise lifestyle intervention guidance to patients.
2. FMT/ placebo intervention-patients will receive three interventions every two weeks.

   Four donors of any gender will be recruited for this study. Patients will receive 200ml FMT from donors with the same gender or receive the same amount of placebo FMT. FMT will be packaged in a 50ml sterile syringe or in an enema bag/surgical nutrition bag, the outer package of which will be affixed with the unique identifiable bar code label generated according to the biological specimen bank of the Department of Laboratory Medicine. The placebo FMT will be mainly composed of normal saline and glycerin and will be packaged in the same way as FMT.

   The night before receiving FMT or placebo FMT via nasointestinal tube, patients will go through proton pump inhibitors(oral 20mg esomeprazole or 40mg omeprazole). The end of the nasointestinal tube should reach at least the patient's duodenum, or reach the patient's jejunum if the patient cooperate. To prevent aspiration, the patient's upper body must maintain an upright posture of 45 degrees for 4 hours after the infusion.

   Before the first intervention, information about drug combination, vital signs, physical examination, BMI, body composition analysis and adverse events of patients will be collected, and advice of diet and lifestyle will be given to patients.

   Before the second intervention and before the third intervention, information about drug combination, vital signs, physical examination, BMI, renal function, liver function, blood fat, fasting blood glucose/C-peptide/insulin, body composition analysis and adverse events of patients will be collected, and advice of diet and lifestyle will be given to patients.
3. Follow-up meetings - total follow up of 6 weeks after FMT/placebo intervention. Meetings will occur 2 weeks and 6 weeks after the third intervention.

During every follow-up meeting, information about drug combination, vital signs, physical examination, BMI, inflammatory biomarkers, renal function, liver function, blood fat, HbAlc, fasting blood glucose/C-peptide/insulin, 2-hour postprandial blood glucose/C-peptide/insulin, body composition analysis and adverse events of patients will be collected, and advice of diet and lifestyle will be given to patients. In the second follow-up meeting, there will be a fecal metagenomics sequencing and a serum metabonomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of T2DM (≥2 months) according to the dagnostic and typing criteria of Chinese guideline for type 2 diabetes
* Control the blood glucose level through diet or exercise only and never receive any hypoglycemic agent in the last 8 weeks.
* Continuous treatment with insulin and its analogues for no more than 14 days in the last year. (The duration of treatment with insulin and its analogues for gestational diabetes mellitus is not included)
* 7.0%≤HbA1c≤10.0%
* Fasting plasma glucose(FPG)<15mmol/L
* 24kg/m2≤BMI≤35kg/m2
* Give informed consent and agree to receive FMT
* Agree to maintain the same diet and exercise habit during the whole process.

Exclusion Criteria:

1. Diagnosed with T1D, gestational diabetes mellitus(GDM) or other special type of diabetes.

2. The presence of any of the following medical histories or clinical conditions that the investigator believes the risks of participation in the study outweigh the benefits or the treatment of combined conditions that may affect subject compliance or the objectivity of the study outcomes.

1. Patients with gastrointestinal disease(such as Irritable bowel syndrome, inflammatory bowel disease, peptic ulcer, gastrointestinal bleeding history, etc.) or history of gastrointestinal surgery(such as gastrectomy, gastroenterostomy, bowel resection, etc.) and are assessed to be unsuitable to participate in this clinical trial by researchers.
2. Patients with severe diabetic complications (diabetic ketoacidosis, hyperglycemic hyperosmolar condition etc.) in the last 6 months.
3. Patients in unstable condition and need therapy for proliferative diabetic retinopathy or maculopathy, severe diabetic neuropathy, diabetic foot or intermittent claudication in the last 6 months.
4. Patients with severe kidney diseases and liver diseases or systemic diseases of other viscera.
5. History or condition of following heart disease in the last 6 months

   * Decompensated cardiac insufficiency(graded III or IV in NYHA)
   * History of unstable angina, myocardial infarction, coronary artery bypass grafting, or coronary stent implantation
   * Diagnosed with Severe arrhythmias requiring treatment(like long QT syndrome etc.), and assessed to be unsuitable to participate in this clinical trial by researchers
6. Patients with uncontrolled hypertension (systolic blood pressure (SBP) ≥ 160mmHg or diastolic blood pressure (DBP) ≥ 100mmHg at screening time).
7. Diagnosed with hemorrhagic stroke or ischemia stroke in the last 6 months and assessed to be unsuitable to participate in this clinical trial by researchers.
8. History of other severe endocrine system diseases that affect glucose metabolism or body weight, such as multiple endocrine adenomas, acromegaly syndrome, Cushing's syndrome, and hyperthyroidism and assessed to be unsuitable to participate in this clinical trial by researchers.
9. History of malignant tumor in the last 5 years (cured basal cell carcinoma of the skin and carcinoma in situ of the cervix are excluded) or malignant tumor being assessed.
10. Patients who have psychiatric disorders or language disorders or are unable or reluctant to communicate, cooperate and be followed up or may have difficulty completing the study judged by the investigator.
11. Patients with severe infection or trauma or history of major surgery in the last 3 months and assessed to be unsuitable to participate in this clinical trial by researchers.
12. History of substance abuse in the last five years, including repeated and large use of dependent medication which is unrelated to medical purposes (addiction medicine and habitual medicine which can lead to physical and mental dependence are included).
13. HIV, TP and HBsAg positive.
14. Participated in any clinical trials of interventional medication or devices in the last 3 months.
15. Patients with anemia or patients who need regular blood transfusion treatment.

3. Receive any of the following medications or treatments.

1. Self-reported weight changes of more than 5kg or use of medication which may result in weight-gain or weight-loss including diuretic, weight loss medicine and so on in the last 90 days.
2. Use of antibiotics in the last 12 weeks.
3. Patients who have used drugs that may affect blood glucose for more than 1 week in the last 12 weeks, such as oral/intravenous glucocorticoid growth hormone, estrogen/progesterone, high-dose diuretics, antipsychotic drugs, etc. (usage of low-dose diuretics (hydrochlorothiazide < 25mg/d, indapamide ≤1.5mg/d) for antihypertensive purposes are not included).
4. Consumption of food or preparation like yogurt, fermented foods, dietary supplements (fish oil, probiotics, prebiotics, various microorganisms, minerals, nutritional foods or herbal preparations) and so on which can affect the gut microbiota in the last 4 weeks.
5. Previous or planned bariatric surgery.

4. Laboratory results during the screening period meet the following criteria.

1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5 upper limit of normal.
2. Glomerular filtration rate(eGFR)< 60 mL/min/1.73m2 calculated by CKD-EPI.
3. Hemoglobin <100g/L
4. Proteinuria 2+ or above.

5. Patients who have suspected or confirmed history of alcohol or drug abuse.

6. Patients known to be allergic to the FMT or its accessories.

7. Pregnancy, breast-feeding, or plans to become pregnant.

8. Patients who are assessed to be unsuitable to participate in this clinical trial by researchers for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of change in weight compared with baseline. | 12 weeks

SECONDARY OUTCOMES:
The absolute value of change in weight compared with baseline. | 6,12 weeks
Proportion of at least 5% reduction in weight. | 12 weeks
Proportion of at least 10% reduction in weight. | 12 weeks
Proportion of at least 15% reduction in weight. | 12 weeks
Proportion of patients with HbA1c < 7.0%. | 12 weeks
Proportion of patients with HbA1c < 6.5%. | 12 weeks
Change in the level of HbA1c. | 6,12 weeks
Change in FCP (fasting C-peptide) compared with baseline. | 6,12 weeks
Change in FPG (fasting plasma glucose) compared with baseline. | 6,12 weeks
Change in FINS (fasting serum insulin) compared with baseline. | 6,12 weeks
Change in 2h-PPG (Postprandial plasma glucose) compared with baseline. | 6,12 weeks
Change in the level of 2-hour postprandial C-peptide compared with baseline. | 6,12 weeks
Change in the level of 2-hour postprandial serum insulin compared with baseline. | 6,12 weeks
Change in BMI compared with baseline. | 6,12 weeks
Change in waist circumference compared with baseline. | 6,12 weeks
Change in hip circumference compared with baseline. | 6,12 weeks
Change in waist hip ratio compared with baseline. | 6,12 weeks
Change in body fat rate compared with baseline. | 6,12 weeks
Change in visceral fat area compared with baseline. | 6,12 weeks
Change in basal metabolic rate compared with baseline. | 6,12 weeks
Change in TC、TG、HDL and LDL compared with baseline. | 6,12 weeks
Change in Blood pressure parameter (SBP, DBP) compared with baseline. | 6,12 weeks
Change in inflammatory markers (hS-CRP, IL-6) compared with baseline. | 6,12 weeks
Change in gut microbiota composition compared with baseline. | 12 weeks
Change in serum metabolic profile compared with baseline. | 12 weeks
Safety of FMT | 12 weeks
  Rate of adverse events(reflux, aspiration, nausea, vomiting belching, abdominal distension, abdominal pain, diarrhea, constipation, infection, fever etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chen, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China